CLINICAL TRIAL: NCT05638165
Title: Phase 1 Clinical Trial to Evaluate the Safety, Tolerability and Efficacy of NCP112
Brief Title: A Single-center, Randomized, Double-blinded, Placebo-controlled, Phase 1 Clinical Trial to Evaluate the Safety, Tolerability and Efficacy of NCP112
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NovaCell Technology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCP112-101
Record Dates: First submitted 2022-11-25; First posted 2022-12-06 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: A Single-center, Randomized, Double-blinded, Placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort QD, NCP112 Gel 0.05% (Experimental): Single dose of NCP112 Gel 0.05% or Single dose of Placebo
  Interventions: Drug: NCP112
- Cohort BID, NCP112 Gel 0.05% (Experimental): Multiple dose of NCP112 Gel 0.05% or Multiple dose of Placebo
  Interventions: Drug: NCP112

INTERVENTIONS:
Drug: NCP112 — The first two subjects for sentinel dosing are randomly assigned to either the test drug or placebo in a 1:1 ratio. After safety and tolerability were reviewed for sentinel participants up to 24 hours after dosing, the subsequent 7 subjects are randomized to the remaining treatment allocations, with 5 subjects to the test drug and 2 to the placebo.

SUMMARY:
To evaluate safety, tolerability and pharmacokinetics of NCP 112 after single and multiple applications on the skin of healthy male volunteers.

DETAILED DESCRIPTION:
Atopic dermatitis is presented as eczematous lesions. Some rashes, discharge, and blisters appear at the acute stage and skin lesions of lichenification appear as the skin becomes thick and leathery at the chronic stage. If not treated properly, a vicious cycle of inflammation of the immune system and further damage to the skin barrier is produced. In particular, enhanced immune reaction to external environmental stimuli plays a major role in inducing pruritis, an essential feature of atopic dermatitis. Pruritis triggers scratching, which in turn leads to an 'itch-scratch-itch' vicious cycle', resulting in secondary skin changes. Therefore, it is important to break the vicious cycle, which worsens the symptoms by means of an optimal treatment.

NCP112 is a first-in-class drug candidate, with a novel target strategy for atopic dermatitis, different from those of the other currently available drugs; The Investigators believe that NCP112 might show a potential as an effective therapy for atopic dermatitis in animal models. Since the efficacy and safety have not been fully elucidated, new adverse reactions, unidentified from the non-clinical data, could appear later. Provided that NCP112 effectively alleviates atopic dermatitis, an intractable chronic disease, it is presumed that the expected benefits would outweigh the foreseeable risks. In the present trial, safety, including occurrences of adverse drug reactions, was thoroughly observed.

This trial was designed as a single-center, block-randomized, double-blind, placebo-controlled, single and multiple dose-ascending trial in which subjects were allocated to either topical application of NCP112 or placebo (vehicle).

The purpose of the present trial was to primarily access the safety of NCP112, the test drug of the trial, in healthy male adults prior to administer the test drug to the real patients with atopic dermatitis, the proposed indication.

ELIGIBILITY:
Inclusion Criteria:

1. A Subject who received and fully understood detailed explanations about the present clinical trial, and whose written consent to participate in the trial and adhere to the precautions was voluntarily obtained before any screening procedures
2. A healthy Korean male adult of age 19 to 55 years of age, inclusive, on the day of signing the informed consent form
3. A Subject who did not have any clinically significant abnormalities observed in physical examination, clinical laboratory tests, electrocardiography, and medical history at the investigator's discretion during the screening
4. A Subject who was able to communicate in Korean with the investigator and comply with the requirements of the protocol as judged by the investigator

Exclusion Criteria:

1. A subject who had a body mass index (BMI) outside the 18.0 ~ 27.0 kg/m² at screening.
2. A subject who had a systolic blood pressure outside the 90 ~ 140 mmHg at screening; or A subject who had a diastolic blood pressure outside the 60 ~ 90 mmHg at screening
3. QTc interval exceeding 450 ms on a 12-lead electrocardiogram at screening
4. A subject who did not meet the following criteria as to the clinical laboratory tests at screening

   * ALT, AST ≤ upper normal level (ULN)x 2.0
   * Total bilirubin, Serum Creatinine ≤ upper normal level (ULN)x 1.5
   * eGFR ≥ 60 mL/min/1.73m²
5. A subject who has a history of alcohol or drug abuse; or has a positive test result for drug/alcohol abuse at screening
6. At the discretion of the investigator, the condition for the cutaneous application of the IP is not suitable for assessment due to the following reasons

   * Dermatologic diseases
   * Damaged skin area to be assessed not suitable for assessment due to sun burn, excessive tanning, uneven skin tone, tattoo, scar, excessive body hair or freckles
7. A subject who has a known history of any allergic diseases such as atopic/allergic diseases (asthma, urticaria, eczematous dermatitis) and food allergy; or eczema
8. A subject who has a known history of allergy or hypersensitivity to any component of the formulation of the IP or peptide drug
9. A subject who has taken any medicine (prescription and non-prescription drug, oriental herbal medicine, health supplementary food, nutritional Supplements) within 2 weeks of the IP dosing
10. A subject who has participated in any clinical trial and taken any IP within 6 months of the IP dosing

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Having observe the predefined safety events from Day 1(the first day of dosing) until Day 8(the day following the final dose)
  Occurrences of 'dosage limiting' toxicity will evaluate in the subjects included in the Safety Set.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No